CLINICAL TRIAL: NCT01860846
Title: Improvement of Work Productivity and Quality of Life With Anti-TNF Therapies Used in Crohn's Disease in Routine Clinical Practice in Turkey
Brief Title: Anti-Tumor Necrosis Factor (TNF) Treatments, Work Productivity and Quality of Life in Crohn's Disease
Acronym: IDEA
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P13-338
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with moderate to severe Crohn's Disease: Participants for whom the treating physician had recently initiated an anti-Tumor Necrosis Factor (TNF) treatment

SUMMARY:
This multicenter, prospective, post marketing observational study (PMOS) was designed to demonstrate long-term effects of anti-Tumor Necrosis Factor therapies on Work Productivity and Impairment scales in participants with moderate to severe Crohn's Disease (CD) under routine conditions. Secondary objectives of this study were long-term improvement of Quality of Life (QoL), evaluation of improvement of extraintestinal symptoms and comorbidities, and evaluation of safety.

DETAILED DESCRIPTION:
Male or female participants between 18 - 65 years of age with moderate to severe CD for whom the treating physician had recently initiated an anti-TNF treatment were included in this study. Anti-TNF treatments were administered according to the treating physician's decision and applicable product label in Turkey. No interventions were made to the treatment and the participant discontinuance or to the follow-up decisions of the treating physician. Enrolled participants were observed for one year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 18-65 years of age with moderately to severely (Crohn's Disease Activity Index 220-450) active Crohn's Disease with or without fistula formation
* Participants who were able to provide authorization to use and disclose information related to the study
* Proven diagnosis of Crohn's Disease in accordance with international diagnostic criteria such as European Crohn's and Colitis Organization (ECCO) guidelines
* Participants for whom the physician had initiated anti-Tumor Necrosis Factor treatment in accordance with Turkish Ministry of Health regulations and reimbursements

Exclusion Criteria:

* Participants who had a history of any kind of biological therapy and/or anti-Tumor Necrosis Factor treatments for Crohn's Disease or other indications
* Participants who had septic complications (active infection and/or active tuberculosis (TB), undrained abscess)
* Participants who had bowel obstructions and fibrotic strictures
* Participants who had received any investigational drug within 30 days prior to the Visit 1 at baseline
* For any reason, participants who were considered by the investigator to be unsuitable

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Crohn's Disease who at the time of study entry were receiving anti-Tumor Necrosis Factor treatment as prescribed in accordance with Turkish Ministry of Health regulations and reimbursement conditions
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2013-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Gücük, MD, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 106 participants were enrolled in the study and were intended to be followed for 12 months.
Period: Overall Study
Arm/Group | Participants With Moderate to Severe Crohn's Disease
Started | 106
Month 1 | 97
Month 2 | 83
Month 4 | 82
Month 6 | 85
Month 12 | 73
Completed | 73
Not Completed | 33
Not completed — Lost to Follow-up | 33

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Participants With Moderate to Severe Crohn's Disease
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 68
Anti-TNF Treatments [Count of Participants; unit: Participants] — Population: Participants with available data
  Participants
    number analyzed (Participants) | 101
    Adalimumab | 78
    Infliximab | 23

OUTCOME MEASURES:

1. Primary Outcome: Work Productivity and Activity Index (WPAI): Absenteeism
Description: The Work Productivity and Activity Impairment: General Health (WPAI:GH) questionnaire was used to assess impairments in both paid work and unpaid work due to symptoms of Crohn's Disease. The self-administered questionnaire consisted of 6 questions. Question 2 asked participants to indicate the number of hours missed due to health problems in the past 7 days. Question 4 asked participants to indicate the number of hours that they worked in the past 7 days. Absenteeism (work time missed) was defined as the percentage of time absent from work due to health problems in the past week and was calculated by the formula Q2/(Q2 + Q4) × 100%. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: At baseline and 12 months
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Moderate to Severe Crohn's Disease
Number analyzed (Participants) | 67
units on a scale
  Baseline | 38.3 (39.0)
  12 months: number analyzed (Participants) | 33
  12 months | 14.2 (27.0)
Statistical Analysis 1: Comparison: Participants With Moderate to Severe Crohn's Disease; The null hypothesis was set as no difference; Test type: Superiority or Other; p = 0.004, Wilcoxon signed-ranked test — Baseline vs. 12 months

2. Primary Outcome: Work Productivity and Activity Index (WPAI): Presenteeism
Description: The Work Productivity and Activity Impairment: General Health (WPAI:GH) questionnaire was used to assess impairments in both paid work and unpaid work due to symptoms of Crohn's Disease. The self-administered questionnaire consisted of 6 questions. Question 5 asked participants the degree to which their health affected productivity while working in the past 7 days, on a scale ranging from 0 to 10, with 0 indicating that health problems had no effect on their work and 10 indicating that health problems completely prevented the participant from working. Presenteeism (impairment at work) was calculated by the formula (Q5/10) × 100%. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: At baseline and 12 months
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Moderate to Severe Crohn's Disease
Number analyzed (Participants) | 58
units on a scale
  Baseline | 39.8 (31.7)
  12 months: number analyzed (Participants) | 40
  12 months | 21.8 (19.3)
Statistical Analysis 1: Comparison: Participants With Moderate to Severe Crohn's Disease; The null hypothesis was set as no difference; Test type: Superiority or Other; p = 0.022, Wilcoxon signed-ranked test — Baseline vs. 12 Months

3. Primary Outcome: Total Work Productivity Impairment (TWPI)
Description: The Work Productivity and Activity Impairment: General Health (WPAI:GH) self-administered questionnaire was used to assess impairments in work due to symptoms of Crohn's Disease. Q2 asked participants the number of hours missed due to health problems in the past 7 days. Q4 asked participants the number of hours that they worked in the past 7 days. Q5 asked participants the degree to which their health affected productivity while working in the past 7 days, on a scale ranging from 0 (health problems had no effect) to 10 (health problems completely prevented them from working). Total work productivity impairment (TWPI) is the combined absenteeism and presenteeism for employed participants, the percentage of overall work productivity lost due to health problems. TWPI was calculated using the formula Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4)))×(Q5/10)] × 100%. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: At baseline and 12 months
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Moderate to Severe Crohn's Disease
Number analyzed (Participants) | 57
units on a scale
  Baseline | 24.2 (21.2)
  12 months: number analyzed (Participants) | 33
  12 months | 15.7 (16.4)
Statistical Analysis 1: Comparison: Participants With Moderate to Severe Crohn's Disease; The null hypothesis was set as no difference; Test type: Superiority or Other; p = 0.006, Wilcoxon signed-ranked test — Baseline vs. 12 Months

4. Primary Outcome: Total Activity Impairment (TAI)
Description: The Work Productivity and Activity Impairment: General Health (WPAI:GH) questionnaire was used to assess impairments in both paid work and unpaid work due to symptoms of Crohn's Disease. The self-administered questionnaire consisted of 6 questions. Question 6 asked participants to indicate the degree to which their health affected their regular activities in the past 7 days. Total activity impairment is the percent impairment of non-work related activities due to health problems and was calculated with the formula (Q6/10) × 100%. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: At baseline and 12 months
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Moderate to Severe Crohn's Disease
Number analyzed (Participants) | 105
units on a scale
  Baseline | 47.0 (32.0)
  12 months: number analyzed (Participants) | 62
  12 months | 30.0 (27.0)
Statistical Analysis 1: Comparison: Participants With Moderate to Severe Crohn's Disease; The null hypothesis was set as no difference; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-ranked test — Baseline vs. 12 Months

5. Secondary Outcome: Change in Short Form 36 (SF-36) Health Survey Scores
Description: The Short Form 36 (SF-36) Health Survey was used to determine participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Scores on each item were summed and averaged (range = 0 "worst" to 100 "best"). Increases from baseline indicate improvement.
Time Frame: At baseline and 12 months
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Moderate to Severe Crohn's Disease
Number analyzed (Participants) | 105
units on a scale
  Physical Functioning Score (Baseline) | 62.8 (30.1)
  Physical Functioning Score (12 months): number analyzed (Participants) | 61
  Physical Functioning Score (12 months) | 81.2 (21.4)
  Role-Physical Score (Baseline) | 29.3 (39.1)
  Role-Physical Score (12 months): number analyzed (Participants) | 61
  Role-Physical Score (12 months) | 67.2 (41.5)
  Role-Emotional Score (Baseline) | 35.2 (39.2)
  Role-Emotional Score (12 months): number analyzed (Participants) | 61
  Role-Emotional Score (12 months) | 62.8 (43.9)
  Vitality Score (Baseline) | 46.9 (26.9)
  Vitality Score (12 months): number analyzed (Participants) | 61
  Vitality Score (12 months) | 58.6 (20.8)
  Mental Health Score (Baseline) | 53.6 (23.6)
  Mental Health Score (12 months): number analyzed (Participants) | 61
  Mental Health Score (12 months) | 63.0 (16.6)
  Social Functioning Score (Baseline) | 58.6 (27.4)
  Social Functioning Score (12 months): number analyzed (Participants) | 61
  Social Functioning Score (12 months) | 70.3 (22.6)
  Bodily Pain Score (Baseline) | 51.9 (30.0)
  Bodily Pain Score (12 months): number analyzed (Participants) | 61
  Bodily Pain Score (12 months) | 73.0 (23.7)
  General Health Score (Baseline) | 44.8 (22.2)
  General Health Score (12 months): number analyzed (Participants) | 61
  General Health Score (12 months) | 54.9 (19.7)
Statistical Analysis 1: Comparison: Participants With Moderate to Severe Crohn's Disease; Physical Functioning Scores: the null hypothesis was set as no difference; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-ranked test — Baseline vs. 12 Months
Statistical Analysis 2: Comparison: Participants With Moderate to Severe Crohn's Disease; Role-Physical Scores: the null hypothesis was set as no difference; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-ranked test — Baseline vs. 12 Months
Statistical Analysis 3: Comparison: Participants With Moderate to Severe Crohn's Disease; Role-Emotional Scores: the null hypothesis was set as no difference; Test type: Superiority or Other; p = 0.001, Wilcoxon signed-ranked test — Baseline vs. 12 Months
Statistical Analysis 4: Comparison: Participants With Moderate to Severe Crohn's Disease; Vitality Scores: the null hypothesis was set as no difference; Test type: Superiority or Other; p = 0.019, Wilcoxon signed-ranked test — Baseline vs. 12 Months
Statistical Analysis 5: Comparison: Participants With Moderate to Severe Crohn's Disease; Mental Health Scores: the null hypothesis was set as no difference; Test type: Superiority or Other; p = 0.017, Wilcoxon signed-ranked test — Baseline vs. 12 Months
Statistical Analysis 6: Comparison: Participants With Moderate to Severe Crohn's Disease; Social Functioning Scores: the null hypothesis was set as no difference; Test type: Superiority or Other; p = 0.007, Wilcoxon signed-ranked test — Baseline vs. 12 Months
Statistical Analysis 7: Comparison: Participants With Moderate to Severe Crohn's Disease; Bodily Pain Scores: the null hypothesis was set as no difference; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-ranked test — Baseline vs. 12 Months
Statistical Analysis 8: Comparison: Participants With Moderate to Severe Crohn's Disease; General Health Scores: the null hypothesis was set as no difference; Test type: Superiority or Other; p = 0.005, Wilcoxon signed-ranked test — Baseline vs. 12 Months

6. Secondary Outcome: Change in Inflammatory Bowel Disease Questionnaire (IBDQ) Scores
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) is a 32-item self-administered questionnaire to measure health-related quality of life in adults with Crohn's Disease. The 32 items are grouped into subscales: bowel-related symptoms (10 items), systemic symptoms (5 items), social function (5 items), and emotional function (12 items). Responses to each item within each subscale range from 1 (significant impairment) to 7 (no impairment), and mean scores ranging from 1 to 7 are calculated for each subscale. Higher scores indicate a better quality of life.
Time Frame: At baseline and 12 months
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Moderate to Severe Crohn's Disease
Number analyzed (Participants) | 105
units on a scale
  Bowel-related Symptoms Score (Baseline) | 4.5 (1.1)
  Bowel-related Symptoms Score (12 months): number analyzed (Participants) | 64
  Bowel-related Symptoms Score (12 months) | 5.2 (1.1)
  Systemic Symptoms Score (Baseline) | 3.8 (1.4)
  Systemic Symptoms Score (12 months): number analyzed (Participants) | 64
  Systemic Symptoms Score (12 months) | 4.9 (1.1)
  Emotional Function Score (Baseline) | 4.0 (1.1)
  Emotional Function Score (12 months): number analyzed (Participants) | 64
  Emotional Function Score (12 months) | 4.7 (1.0)
  Social Function Score (Baseline) | 4.3 (1.5)
  Social Function Score (12 months): number analyzed (Participants) | 64
  Social Function Score (12 months) | 5.3 (1.5)
Statistical Analysis 1: Comparison: Participants With Moderate to Severe Crohn's Disease; Bowel-related Symptoms Scores: The null hypothesis was set as no difference; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-ranked test — Baseline vs. 12 Months
Statistical Analysis 2: Comparison: Participants With Moderate to Severe Crohn's Disease; Systemic Symptoms Scores:The null hypothesis was set as no difference; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-ranked test — Baseline vs. 12 Months
Statistical Analysis 3: Comparison: Participants With Moderate to Severe Crohn's Disease; Emotional Function Scores: the null hypothesis was set as no difference; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-ranked test — Baseline vs. 12 Months
Statistical Analysis 4: Comparison: Participants With Moderate to Severe Crohn's Disease; Social Function Scores: The null hypothesis was set as no difference; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-ranked test — Baseline vs. 12 Months

7. Secondary Outcome: Change in Extra-intestinal Symptoms
Description: Extra-intestinal manifestations of Crohn's Disease (skeletal system [bones and muscle], dermatological [skin], hepatobiliary system [liver, gall bladder, and bile ducts], ocular [eyes] and oral [mouth]) were documented by the study investigators at each visit.
Time Frame: At baseline and 12 months
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Moderate to Severe Crohn's Disease
Number analyzed (Participants) | 106
Participants
  Skeletal symptoms present (Baseline) | 20
  Skeletal symptoms present (12 months): number analyzed (Participants) | 73
  Skeletal symptoms present (12 months) | 8
  Dermatological symptoms present (Baseline) | 7
  Dermatological symptoms present (12 months): number analyzed (Participants) | 73
  Dermatological symptoms present (12 months) | 3
  Hepatobiliary symptoms present (Baseline) | 0
  Hepatobiliary symptoms present (12 months): number analyzed (Participants) | 73
  Hepatobiliary symptoms present (12 months) | 0
  Ocular symptoms present (Baseline) | 1
  Ocular symptoms present (12 months): number analyzed (Participants) | 73
  Ocular symptoms present (12 months) | 0
  Oral symptoms present (Baseline) | 4
  Oral symptoms present (12 months): number analyzed (Participants) | 73
  Oral symptoms present (12 months) | 0

8. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: A serious adverse event was defined as any untoward medical occurrence in a clinical investigation participant that met at least 1 of the following criteria: death, life-threatening, hospitalization or prolongation of hospitalization, congenital anomaly, persistent or significant disability/incapacity, important medical event requiring medical or surgical intervention to prevent serious outcome, elective or spontaneous abortion.
Time Frame: From the time of informed consent until 30 days or 5 half-lives following the last dose, up to 62 weeks
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Moderate to Severe Crohn's Disease
Number analyzed (Participants) | 106
Participants | 2

ADVERSE EVENTS:
Time Frame: From the time of informed consent until 30 days or 5 half-lives following the last dose, up to 62 weeks
Description: Nonserious adverse events were not collected for this study.
Arm/Group | Participants With Moderate to Severe Crohn's Disease
Serious Adverse Events (participants affected / at risk) | 2/106
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Moderate to Severe Crohn's Disease (N=106)
Abdominal abscess (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
Participants lost to follow-up were not replaced. Participant selection bias and lower number of participants completing questionnaires at later study visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.